CLINICAL TRIAL: NCT07086573
Title: The Effect of Algae Oil Supplements on Functional Immune Response and Bioavailability of Lipids in Blood, a Pilot Study
Acronym: ALG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maartje van den Belt (Other)
Collaborators: Nutricia Research (Industry); Fermentalg (Unknown); Microalgas Oleas de México, S.A. de C.V. (Unknown); Utrecht University (Other)
Responsible Party: Sponsor-Investigator, Maartje van den Belt, Researcher Food, Health & Consumer research, Wageningen University and Research
Organization: Wageningen University and Research (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023-16979
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Functional Immune Response; Postprandial Bioavailability DHA; Fatty Acid Metabolism
Keywords: Immune function; DHA bioavailability; ALG study; Algae oil; Omega-3
MeSH Terms: interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: The study is a randomized, crossover, double-blind, controlled study of 7 weeks with 3 study arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fish oil (control) (Active Comparator): Tuna oil
  Interventions: Dietary Supplement: Fish oil (control)
- Algae oil supplement 1 (Experimental): Algae oil 1
  Interventions: Dietary Supplement: Algae oil 1
- Algae oil supplement 2 (Experimental): Algae oil 2
  Interventions: Dietary Supplement: Algae oil 2

INTERVENTIONS:
Dietary Supplement: Algae oil 1 — DHA Origins 550-Y oil (Fermentalg)
  Arms: Algae oil supplement 1
Dietary Supplement: Algae oil 2 — Oleo H-02 (Microalgas)
  Arms: Algae oil supplement 2
Dietary Supplement: Fish oil (control) — Tuna oil
  Arms: Fish oil (control)

SUMMARY:
In this explorative study we will investigate whether two sustainable oil supplements yield equivalent results to fish oil supplements in terms of postprandial immune response, among elderly adults, after standardization of the quantity of DHA among the oils. Results on the bioavailability of DHA from different oil supplements will help determine whether differences in DHA bioavailability lead to differences in immune function. Additionally, we will investigate postprandial inflammatory markers. The outcomes of this exploratorive study will provide insight into the variation between individuals and potential effect sizes, and will aim to conduct more targeted follow-up studies on the effects of algae oils on immune function.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy men and women;
* Age ≥ 50 years
* Body mass index (BMI) ≥18.5 and ≤30 kg/m2;
* Having veins suitable for blood sampling via a catheter (judged by study nurse/ medical doctor);
* Willing to refrain from fish, fish oil, and products with added omega-3 starting from 2 weeks prior to first postprandial test day.
* Willing to keep a stable dietary pattern throughout the study

Exclusion Criteria:

* Having a disease that may interfere with the outcomes of this study, such as a known metabolic, gastrointestinal, inflammatory or chronic disease (such as anaemia, diabetes, hepatitis, cardiovascular disease), as judged by the medical investigator;
* Having a history of medical or surgical events that may significantly affect the study outcome, including: inflammatory bowel disease, hepatitis, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer;
* Use of medication that may interfere with the study outcomes, including gastric acid inhibitors or laxatives, as judged by the medical supervisor.
* Anaemia (Haemoglobin (Hb) values <7.5 mmol/L for women and <8.5 mmol/L for men), as assessed by finger prick blood during screening visit;
* Having swallowing problems with capsules;
* Allergic for fish or shellfish;
* Recent blood donation (<1 month prior to test day 1 of the study) or not willing to stop donation during and 1 month after the study;
* Average alcohol intake >21 (women) or >28 (men) glasses of alcoholic beverages per week;
* Reported weight loss or weight gain of more than 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period;
* Reported to follow or having planned a slimming or medically prescribed diet;
* Use of drugs;
* Current smokers, or stopped smoking in the last 3 months before study start;
* Insufficient proficiency in Dutch to understand information brochure and questionnaires;
* Participation in any clinical trial including blood sampling and/or administration of sub-stances up to 30 days before test day 1 of this study and during the study period;
* Being an employee of the department Food, Health & Consumer Research Wageningen Food & Biobased Research or Food Quality and Design of Wageningen University.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Functional immune response | Baseline (0 hours)
  Measured in isolated PBMCs by calculating the ratio of pro- and anti-inflammatory markers after ex vivo stimulation with LPS and measurement of the cytokine response. The following markers will be measured: pro inflammatory (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5), anti-inflammatory (IL-4 and IL-10).
Functional immune response | 4 hours postprandial
  Measured in isolated PBMCs by calculating the ratio of pro- and anti-inflammatory markers after ex vivo stimulation with LPS and measurement of the cytokine response. The following markers will be measured: pro inflammatory (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5), anti-inflammatory (IL-4 and IL-10).
Functional immune response | 8 hours postprandial
  Measured in isolated PBMCs by calculating the ratio of pro- and anti-inflammatory markers after ex vivo stimulation with LPS and measurement of the cytokine response. The following markers will be measured: pro inflammatory (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5), anti-inflammatory (IL-4 and IL-10).
Functional immune response | 1 week after exposure to the oil
  Measured in isolated PBMCs by calculating the ratio of pro- and anti-inflammatory markers after ex vivo stimulation with LPS and measurement of the cytokine response. The following markers will be measured: pro inflammatory (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5), anti-inflammatory (IL-4 and IL-10).

SECONDARY OUTCOMES:
Plasma DHA levels | Baseline (0 hours)
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 1 hour postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 2 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 3 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 4 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 5 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 6 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 7 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Plasma DHA levels | 8 hours postprandial
  Measured in venous blood samples. DHA will be determined by gas chromatography.
Fatty acid levels in plasma and PBMCs | Baseline (0 hours)
  Measured in plasma and PBMCs, fatty acids will be determined by gas chromatography.
Fatty acid levels in plasma and PBMCs | 1 week after exposure to the oil
  Measured in plasma and PBMCs, fatty acids will be determined by gas chromatography.

OTHER OUTCOMES:
Plasma EPA levels | Baseline (0 hours)
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 1 hour postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 2 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 3 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 4 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 5 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 6 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 7 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Plasma EPA levels | 8 hours postprandial
  Measured in venous blood samples. Plasma EPA will be determined by gas chromatography
Functional immune response in plasma | Baseline
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 1 hour postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 2 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 3 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 4 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 5 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 6 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 7 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Functional immune response in plasma | 8 hours postprandial
  The ratio of pro (PGE2, IL-1β, IL-6, IL-8, IFNg, TNFα, CCL2 and CCL5) and anti-inflammatory markers (IL-4 and IL-10) will be determined using ELISA kits or a custom LegendPlex.
Oxylipin levels in plasma | Baseline (0 hours)
  Oxylipin levels will be determined by LC-MS/MS after solid phase extraction
Oxylipin levels in plasma | 4 hours postprandial
  Oxylipin levels will be determined by LC-MS/MS after solid phase extraction
Oxylipin levels in plasma | 8 hours postprandial
  Oxylipin levels will be determined by LC-MS/MS after solid phase extraction
Oxylipin levels in plasma | 1 week after exposure to the oil
  Oxylipin levels will be determined by LC-MS/MS after solid phase extraction
Fatty acid levels in cell membranes of erythrocytes | Baseline (0 hours)
  Fatty acid levels in cell membranes of erythrocytes will be determined by gas chromatography
Fatty acid levels in cell membranes of erythrocytes | 1 week after exposure to the oil
  Fatty acid levels in cell membranes of erythrocytes will be determined by gas chromatography
Gastrointestinal complaints | Baseline (0 hours)
  Abdominal pain, bloating, flatulence, gastric acid, nausea, diarrhea on a VAS scale (0-10)
Gastrointestinal complaints | 4 hours postprandial
  Abdominal pain, bloating, flatulence, gastric acid, nausea, diarrhea on a VAS scale (0-10)
Gastrointestinal complaints | 8 hours postprandial
  Abdominal pain, bloating, flatulence, gastric acid, nausea, diarrhea on a VAS scale (0-10)
Gastrointestinal complaints | 12 hours postprandial
  Abdominal pain, bloating, flatulence, gastric acid, nausea, diarrhea on a VAS scale (0-10)
Gastrointestinal complaints | 1 week after exposure to the oil
  Abdominal pain, bloating, flatulence, gastric acid, nausea, diarrhea on a VAS scale (0-10)
Short term well-being | Baseline (0 hours)
  Short-term well-being assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short term well-being | 4 hours postprandial
  Short-term well-being assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short term well-being | 8 hours postprandial
  Short-term well-being assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short term well-being | 12 hours postprandial
  Short-term well-being assessed by the Multidimensional Mood Questionnaire (MDMQ)
Short term well-being | 1 week after exposure to the oil
  Short-term well-being assessed by the Multidimensional Mood Questionnaire (MDMQ)

CONTACTS AND LOCATIONS:
Overall Officials: Maartje van den Belt, MSc, Principal Investigator — Wageningen Food and Biobased Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Since study participants did not give consent to share data with other parties.